CLINICAL TRIAL: NCT00872235
Title: An Open Label, Balanced, Randomised, Two-Treatment, Four-Period, Two-Sequence, Single-Dose, Crossover, Fully Replicated Bioavailability Study on Fixed-Dose Combination of Quinapril 20 mg and Hydrochlorothiazide 25 mg Tablets of OHM Laboratories Inc.(Division of Ranbaxy Laboratories Limited) With Accuretic 20-25 mg Tablets (Fixed Dose Combination of Quinapril 20 mg and Hydrochlorothiazide 25 mg) of Parke-Davis (Division of Pfizer Inc.) in Healthy, Adult, Human, Male Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Quinapril Hydrochloride 20 mg and Hydrochlorothiazide 25 mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CPU-M-024/QUINH-45/05
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Healthy
Keywords: Bioequivalence fixed-dose combination of quinapril 20 mg and hydrochlorothiazide 25 mg tablets
MeSH Terms: interventions — Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): fixed-dose combination of quinapril 20 mg and hydrochlorothiazide 25 mg tablets of OHM Laboratories Inc.(division of Ranbaxy Laboratories Limited)
  Interventions: Drug: fixed-dose combination of quinapril 20 mg and hydrochlorothiazide 25 mg tablets
- 2 (Active Comparator): Accuretic tablets (fixed dose combination of quinapril 20 mg and hydrochlorothiazide 25 mg)
  Interventions: Drug: fixed-dose combination of quinapril 20 mg and hydrochlorothiazide 25 mg tablets
- 3 (Experimental): fixed-dose combination of quinapril 20 mg and hydrochlorothiazide 25 mg tablets of OHM Laboratories Inc.(division of Ranbaxy Laboratories Limited)
  Interventions: Drug: fixed-dose combination of quinapril 20 mg and hydrochlorothiazide 25 mg tablets
- 4 (Active Comparator): Accuretic tablets (fixed dose combination of quinapril 20 mg and hydrochlorothiazide 25 mg)
  Interventions: Drug: fixed-dose combination of quinapril 20 mg and hydrochlorothiazide 25 mg tablets

INTERVENTIONS:
Drug: fixed-dose combination of quinapril 20 mg and hydrochlorothiazide 25 mg tablets

SUMMARY:
This open-label, balanced, randomized, two-treatment, four-period, two-sequence, single dose, crossover fully replicated study was conducted on fixed-dose combination of quinapril 20 mg and hydrochlorothiazide 25 mg tablets of OHM Laboratories Inc. (division of Ranbaxy Laboratories Limited) and Accuretic 20-25 mg tablets of Parke-Davis (division of Pfizer Inc.) in healthy, adult, human, male, subjects under fed conditions.

DETAILED DESCRIPTION:
The subjects received a single oral dose of either Test or Reference product, containing fixed-dose combination of Quinapril 20 mg and Hydrochlorothiazide 25 mg after an overnight fast of at least 10 hours. The study drug was administered as per the SAS generated Randomization Code, 30 minutes after serving of a high-fat high-calorie breakfast under supervision of a trained Medical Officer in each period.Blood samples were collected predose and at intervals over 72 hours after each dose. A 7-day interval was maintained between each dosing in the Study Periods I-IV.

During the course of the study safety parameters assessed were vital signs, physical examination, medical history, clinical laboratory safety tests (hematology, biochemical parameters and urine analysis) at base line. Laboratory parameters of hematology and biochemistry were repeated and sodium & potassium levels were estimated at the 24 hours post dose of the last period of the study.

A total of 40 subjects were randomized to receive fixed-dose combination of quinapril 20 mg and hydrochlorothiazide 25 mg tablets and 37 subjects completed all the four periods of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be in the age range of 18-45 years.
2. Be neither overweight nor underweight for his/her height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
3. Have voluntarily given written informed consent to participate in this study.
4. Be of normal health as determined by medical history and physical examination of the subjects performed within 14 days prior to the commencement of the study.

Exclusion Criteria:

1. History of allergy to quinapril, hydrochlorothiazide, sulfonamide derived drugs or related ACE inhibitors.
2. History of anuria, gout or dry cough.
3. History of diarrhea or vomiting in the last one week.
4. Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
5. Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
6. Presence of values, which are significantly different from normal, reference ranges (as defined in Appendix 5) and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
7. Positive for urinary screen testing of drugs of abuse (opiates or cannabinoids).
8. Presence of values, which are significantly different from normal, reference ranges (as defined in Appendix 5) and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
9. Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), glucose (positive) or protein (positive).
10. Clinically abnormal ECG or Chest X-ray.
11. History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes, glaucoma or angioedema due to any cause.
12. History of any psychiatric illness which may impair the ability to provide written informed consent.
13. Regular smokers who smoke more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
14. History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or have difficulty in abstaining for the duration of each study period.
15. Use of any enzyme modifying drugs within 30 days prior to Day 1 of this study.
16. Participation in any clinical trial within 12 weeks preceding Day 1 of this study.
17. A haemoglobin concentration of less than 7 % of lower limit of reference range e.g. 13 gm % for reference range of 14-18 gm at screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2005-06; Primary Completion 2005-07 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence evaluation of Quinapril hydrochloride 20 mg and Hydrochlorothiazide 25 mg tablets under fed conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Ranbaxy CPU, New Delhi, New Delhi, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html